CLINICAL TRIAL: NCT07146282
Title: Vitamin K Antagonist in Rheumatic Heart Disease Patients With Mechanical Heart Valves: Our Current Status
Acronym: VKA and RHD
Status: Not yet recruiting | Type: Observational
Sponsor: Ahmed Hassan Rostom Ibrahim (Other)
Responsible Party: Sponsor-Investigator, Ahmed Hassan Rostom Ibrahim, principal investigator, Assiut University
Organization: Assiut University (Other)
Other Study IDs: VKA in RHD current status
Record Dates: First submitted 2025-08-04; First posted 2025-08-28 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Rheumatic Heart Disease
MeSH Terms: conditions — Rheumatic Heart Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
VKA in RHD patients with MHV: our current status

DETAILED DESCRIPTION:
Vitamin K Antagonist in Rheumatic heart disease patients with mechanical heart valves: Our Current Status

ELIGIBILITY:
Inclusion Criteria:

* Confirmed presence of a mechanical heart valve.
* Aged ≥18 years

Exclusion Criteria:

* Pregnancy.
* Active bleeding disorders.
* Severe liver/kidney disease (if affecting anticoagulation).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Data collection: Data will be collected directly by the researcher and will be reviewed by the supervising team to ensure accuracy and consistency. The data collection process will involve recording INR observation , clinical evaluations Each participant will have their data entered into a secure database for further analysis.
Sampling Method: Non-Probability Sample
Enrollment: 165 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2027-09 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Time in therapeutic range (TTR) for warfarin. | Baseline
  TTR status will be calculated using the most recent INR value and patient records to determine whether INR is within the target therapeutic range (2.0-3.5) at the time of data collection.
2. Correlation Between TTR and Patient-Specific Factors | Baseline
  Assesses the relationship between INR control and factors such as age, comorbidities, adherence, vitamin K intake, and medication use based on data collected at the single study visit.

SECONDARY OUTCOMES:
1. Number of Participants With Reported Bleeding Events (Major or Minor) | Baseline
  Presence or absence of self-reported or documented major/minor bleeding events prior to or at the time of data collection.
Number of Participants With Thromboembolic Events | Baseline
  History of stroke, valve thrombosis, or systemic embolism collected from medical records or patient report during the study visit.
Rate of Patient Adherence to Warfarin Therapy | Baseline
  Adherence assessed via patient self-report and/or pill count at the single study visit.

CONTACTS AND LOCATIONS:
Overall Officials: Hamdy Shams Mohamed, Principal Investigator; Tarek hameed Nageeb, Principal Investigator

REFERENCES:
- [Background] Watkins DA, Johnson CO, Colquhoun SM, Karthikeyan G, Beaton A, Bukhman G, Forouzanfar MH, Longenecker CT, Mayosi BM, Mensah GA, Nascimento BR, Ribeiro ALP, Sable CA, Steer AC, Naghavi M, Mokdad AH, Murray CJL, Vos T, Carapetis JR, Roth GA. Global, Regional, and National Burden of Rheumatic Heart Disease, 1990-2015. N Engl J Med. 2017 Aug 24;377(8):713-722. doi: 10.1056/NEJMoa1603693. PMID 28834488
- [Background] Beckmann A, Meyer R, Lewandowski J, Markewitz A, Blassfeld D, Boning A. German Heart Surgery Report 2022: The Annual Updated Registry of the German Society for Thoracic and Cardiovascular Surgery. Thorac Cardiovasc Surg. 2023 Aug;71(5):340-355. doi: 10.1055/s-0043-1769597. Epub 2023 Jun 16. PMID 37327912
- [Background] El-Hamamsy I, Toyoda N, Itagaki S, Stelzer P, Varghese R, Williams EE, Erogova N, Adams DH. Propensity-Matched Comparison of the Ross Procedure and Prosthetic Aortic Valve Replacement in Adults. J Am Coll Cardiol. 2022 Mar 1;79(8):805-815. doi: 10.1016/j.jacc.2021.11.057. PMID 35210036
- [Background] Zilla P, Human P, Pennel T. Mechanical valve replacement for patients with rheumatic heart disease: the reality of INR control in Africa and beyond. Front Cardiovasc Med. 2024 Feb 9;11:1347838. doi: 10.3389/fcvm.2024.1347838. eCollection 2024. PMID 38404722
- See also: Related Info — https://pmc.ncbi.nlm.nih.gov/articles/PMC10884232/